CLINICAL TRIAL: NCT00049374
Title: A Phase II Study Of Genasense In Combination With Thalidomide And Dexamethasone In Relapsed And Refractory Multiple Myeloma
Brief Title: Oblimersen, Thalidomide, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258058; MSGCC-210421; NCI-5824
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — oblimersen; Dexamethasone; Thalidomide

INTERVENTIONS:
Biological: oblimersen sodium
Drug: dexamethasone
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may slow the growth of cancer cells. Oblimersen may increase the effectiveness of thalidomide and dexamethasone by making cancer cells more sensitive to the drugs.

PURPOSE: Phase II trial to study the effectiveness of combining thalidomide and dexamethasone with oblimersen in treating patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical efficacy of oblimersen, thalidomide, and dexamethasone, in terms of complete and partial response rates, in patients with relapsed or refractory multiple myeloma.
* Determine the time to progression and duration of response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Correlate disease response (clinical outcome) with changes in Bcl-2 levels in patients treated with this regimen.
* Determine the disease-free and overall survival of patients treated with this regimen.

OUTLINE: Patients receive induction therapy comprising oblimersen IV continuously on days 1-7, 22-28, and 43-49, oral dexamethasone on days 4-7, 25-28, and 46-49, and oral thalidomide daily beginning on day 4. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients with stable disease after induction therapy receive maintenance therapy comprising oblimersen IV continuously on days 1-7, oral dexamethasone on days 4-7, and oral thalidomide daily. Courses repeat every 35 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 10-46 patients will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and clinically confirmed multiple myeloma

  * Relapsed and/or refractory after chemotherapy or transplantation

    * Patients with prior allogeneic transplantation must not have evidence of active graft-vs-host disease requiring immune suppression
* Measurable disease defined by quantitative immune globulin levels in serum and/or urine and bone marrow plasmacytosis

  * Patients with nonsecretory disease are eligible provided at least 1 plasmacytoma lesion is accurately measurable by MRI or CT scan
* No known CNS involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 50,000/mm^3* NOTE: *Unless secondary to bone marrow plasmacytosis (more than 80% involvement)

Hepatic

* Bilirubin less than 2 times normal
* AST/ALT no greater than 3 times upper limit of normal

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Seizures allowed if under adequate control
* No severe skin reactions from prior thalidomide
* No prior allergic reactions attributed to agents used in this study
* No sensory or motor neuropathy grade II or greater
* No other uncontrolled concurrent illness that would preclude study therapy
* No ongoing or active infection
* No psychiatric illness or social situations that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception for 1 month before, during, and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Chemotherapy
* At least 6 weeks since prior thalidomide

Chemotherapy

* See Disease Characteristics
* No more than 4 prior chemotherapy regimens, including autologous and/or allogeneic stem cell transplantation regimens
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Concurrent continuous steroids allowed for chronic treatment of disorders other than myeloma

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior oblimersen
* No other concurrent anticancer therapies or investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Complete and partial remission

SECONDARY OUTCOMES:
Relationship between molecular and clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Z. Badros, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York

REFERENCES:
- [Result] Badros AZ, Goloubeva O, Rapoport AP, Ratterree B, Gahres N, Meisenberg B, Takebe N, Heyman M, Zwiebel J, Streicher H, Gocke CD, Tomic D, Flaws JA, Zhang B, Fenton RG. Phase II study of G3139, a Bcl-2 antisense oligonucleotide, in combination with dexamethasone and thalidomide in relapsed multiple myeloma patients. J Clin Oncol. 2005 Jun 20;23(18):4089-99. doi: 10.1200/JCO.2005.14.381. Epub 2005 May 2. PMID 15867202